CLINICAL TRIAL: NCT06549985
Title: Interdisciplinary Group Care for the Treatment of Endometriosis-associated Pain: the Peer Empowered Endometriosis Pain Support (PEEPS) Pilot Randomized Controlled Trial
Brief Title: Interdisciplinary Group Care for the Treatment of Endometriosis-associated Pain
Acronym: PEEPS RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202402082
Record Dates: First submitted 2024-08-05; First posted 2024-08-12 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Endometriosis; Pelvic Pain
Keywords: Group care; Integrative care; Pelvic floor physical therapy; Mindfulness; Patient-centered outcomes
MeSH Terms: conditions — Endometriosis; Pelvic Pain | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer Empowered Endometriosis Pain Support (PEEPS) (Experimental): Participants in this arm will receive PEEPS plus usual care. PEEPS is comprised of eight weekly two-hour sessions delivered to groups of 6-10 participants. The sessions provide education on endometriosis, mindfulness, yoga, nutrition, and strategies to cope with chronic pain. Participants additionally receive peer and clinician support.
  Interventions: Behavioral: PEEPS
- Education (Active Comparator): Participants in this arm will receive an educational handout providing the basics of endometriosis pathophysiology, diagnosis, and treatment plus usual care
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: PEEPS — Participants will participate in the PEEPS program in addition to usual care.
  Arms: Peer Empowered Endometriosis Pain Support (PEEPS)
Behavioral: Education — Participants will receive an educational handout on endometriosis in addition to usual care.
  Arms: Education

SUMMARY:
The goal of this clinical trial is to determine if Peer Empowered Endometriosis Pain Support (PEEPS), an 8-week interdisciplinary, integrative group care program, decreases pain interference in participants with endometriosis-associated chronic pelvic pain between the ages 18 and 48. The main question we aim to answer is:

Is PEEPS more effective than Education in decreasing pain interference?

Researchers will compare people receiving PEEPS plus usual care to those receiving Education plus usual care to see if people participating in PEEPS demonstrate improvements in pain, physical function, and quality of life.

Participants will:

* Complete baseline quality of life surveys
* Participate in an 8-session group care program
* Provide feedback on each session and the program globally
* Complete follow up quality of life surveys at PEEPS completion, 6- and 12-months post-completion.
* A sub-set will complete semi-structured interviews or focus groups about the experience of participating in PEEPS

ELIGIBILITY:
Inclusion Criteria:

* Age 18-48 years
* Operative confirmation of endometriosis
* Chronic pelvic pain (pain perceived to originate from the pelvis, not exclusively during menses, lasting ≥6 months)
* No plan to have surgery before or during the PEEPS cohort
* Able to attend at least six of the eight 2-hour weekly sessions on the Washington University campus
* Comfort reading and speaking English as groups and materials are in English

Exclusion Criteria:

* Currently pregnant
* Severe physical impairment (limiting yoga participation)
* History of hip or spine surgery given increased risk of harm and need for extensive activity modification
* Current or history of psychiatric disorder with psychosis in order to minimize risk of adverse mental health effects to participants
* Opioid use ≥ 5 days in the past 3 months, other than for the 6-week post-operative period
* History of surgical removal of bilateral ovaries

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Patient Reported Outcomes Measurement Information System (PROMIS) pain interference Short Form (SF) 8a | Baseline, immediately after the intervention
  Validated, 8-question survey that assesses pain interference in daily activities

OTHER OUTCOMES:
PROMIS pain interference SF 8a | Baseline, 6- and 12-months after the intervention
  Validated, 8-question survey that assesses pain interference in daily activities
PROMIS pain intensity | Baseline, immediately after the intervention, 6- and 12-months after the intervention
  Validated, 3-question survey that measures pain intensity on a 1-5 scale over the past 7 days
Endometriosis Health Profile-30 | Baseline, immediately after the intervention, 6- and 12-months after the intervention
  Validated, 30-question endometriosis-related quality of life measure
PROMIS Physical Function SF10a | Baseline, immediately after the intervention, 6- and 12-months after the intervention
  Validated, 10-questions survey that measures physical function such as walking, carrying groceries, and other activities of daily living
PROMIS Anxiety SF7a | Baseline, immediately after the intervention, 6- and 12-months after the intervention
  Validated, 7-question survey that measures anxiety in past 7 days
PROMIS Depression SF8b | Baseline, immediately after the intervention, 6- and 12-months after the intervention
  Validated, 8-question survey that measures depression in past 7 days
Patient global impression of change | Immediately after the intervention, 6- and 12-months after the intervention
  Validated, 1-question survey on impression of change over time

CONTACTS AND LOCATIONS:
Overall Officials: Whitney Ross, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- WashU Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be preserved and shared through Digital Commons@Becker, an institutional repository administered and maintained by the Bernard Becker Medical Library at Washington University in St. Louis. All de-identified clinical, survey, and interview data from this project will be shared via Digital Commons@Becker of sufficient quality to validate and replicate research findings. Data dictionaries and study protocols will also be shared via Digital Commons@Becker.
Supporting Information: Study Protocol
Time Frame: All scientific data generated from this project will be made available no later than the time of an associated publication or 12 months after completion of the final data point, whichever is sooner.
Access Criteria: The human subjects' data shared will be within the Institutional Review Board (IRB) bounds. The human subject data will be de-identified and made available via controlled access to the approved user(s) who signed the Data Use Agreement (DUA) to ensure the requester(s) have a legitimate reason for access, and agree not to attempt re-identification of participants and not to distribute data to unauthorized users.

REFERENCES:
- [Derived] Ross WT, Buday S, Yakel E, Khabele D, Balls-Berry J, As-Sanie S, Colditz G, Baumann AA. Does interdisciplinary group care for the treatment of endometriosis improve pain interference: protocol for a pilot randomised controlled trial at an urban academic medical centre. BMJ Open. 2025 Mar 5;15(3):e097372. doi: 10.1136/bmjopen-2024-097372. PMID 40044193